CLINICAL TRIAL: NCT04857125
Title: Prevention of Delirium After Acute Surgery - Implementation of a Multicomponent Intervention Throughout the Hospitalization
Brief Title: Prevention of Postoperative Delirium After Acute Surgery
Acronym: POD-CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Sine Eriksen, Principal Investigator, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: H-20067775
Record Dates: First submitted 2021-03-04; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Delirium
Keywords: Implementation; Prevention; Multicomponent intervention; Anaesthetics, General; Non-cardiac; Acute surgery; Non-pharmacological intervention; Postoperative care
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded from the groups, when assessing the primary outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent intervention (Active Comparator): Pre-, intra- and postoperative interventions applied using the Fast-IM method.
  Interventions: Other: Patient interventions; Other: Staff education
- Standard care (No Intervention): Patients are receiving standard care.

INTERVENTIONS:
Other: Patient interventions — The multicomponent intervention consists of several elements regarding avoidance of specific pre-medications and optimising the patients condition before surgery (reducing fasting and fluid-fasting time).
  Per-operative focus on using bispectral index (BIS) guided anaesthesia, Total intravenous anaesthesia (TIVA) as first choice, pain-and PONV (postoperative nausea and vomiting) prophylaxis and treatment.
  Postoperative focus on: Reducing indwelling catheters, Fluid (p.o. or IV), Nutrition, Mobilisation, Sleep, Non-pharmacological interventions (Shielding, involving of relatives, orientation, optimizing of senses)
  Arms: Multicomponent intervention
Other: Staff education — Staff will be educated for at least 1-2 hours. Anaesthesiologist and nurse anaesthetists will receive a brush up on the use of bispectral index (BIS) and the intervention elements that are implemented and monitored. Staff in the PACU, as well as staff in the surgery wards, will be educated in postoperative delirium, learning to identify symptoms of delirium and how to use the screening tool CAM.
  Arms: Multicomponent intervention

SUMMARY:
The aim of this trial is to evaluate the implementation and effect of an evidence based, multicomponent intervention on postoperative delirium, when fast implemented throughout the patients stay in hospital before, during and after acute surgery in a risk population, the primary outcome being frequency of patients with positive Confusion Assessment Method (CAM) score.

The hypothesis is that the frequency of postoperative delirium will be reduced after implementation of the preventive interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 or above.
* Patients scheduled for acute abdominal or orthopaedic surgery in general anaesthesia with an expected duration of 30 minutes or more.
* Patients who are scheduled for surgery within 72 hours of hospital admission.
* Patients who are expected to stay in hospital for 24 hours or more.

Exclusion Criteria:

* Patients screened CAM positive before surgery.
* Patients who have already been included in the study
* Patients unable to speak and read Danish.
* Inability to provide consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium identified with the screening tool Confusion Assessment Method (CAM), assessing change from negative to positive score. | During the 5 initial postoperative in-hospital days. Patients are screened twice a day; in the morning (7-10 AM) and in the evening (7-11 PM).
  Patients are screened with the tool Confusion Assessment Method (CAM). A patient will be considered CAM positive, according to the CAM algorithm for diagnosis of delirium that requires the presence of both the first (acute onset and fluctuating course) and the second criteria (inattention) and of either the third (disorganised thinking) or the fourth criterion (altered level of consciousness).

SECONDARY OUTCOMES:
Inadequate emergence identified with the screening tool Confusion Assessment Method (CAM) in the Post-Anaesthesia Care Unit (PACU), assessing change from negative to positive score. | Patients are screened at time of arrival and until discharge from PACU
  Patients are screened with the tool Confusion Assessment Method (CAM) in the Post-Anaesthesia Care Unit (PACU). A patient will be considered CAM positive, according to the CAM algorithm for diagnosis of delirium that requires the presence of both the first (acute onset and fluctuating course) and the second criteria (inattention) and of either the third (disorganised thinking) or the fourth criterion (altered level of consciousness). A positive CAM score at any time during the PACU stay is considered as having "Inadequate emergence", assessing change from negative to positive score.
All-cause mortality within 30 days. | Day 30
  All-cause mortality
Length of postoperative stay (LOS). | Day 30
  Length of postoperative stay in hospital
Length of stay in the Post-Anaesthesia Care Unit (PACU) after surgery. | Day 30
  Length of stay in the Post-Anaesthesia Care Unit (PACU) after surgery after surgery will be assessed.
Number of participants who are readmitted to hospital within 30 days. | Day 30
  Re-admissions are defined as an acute admission which takes place between 4 hours and 30 days after discharge from hospital. The readmission indicator is non-specific, as all readmissions are included, regardless of which hospital the readmission takes place and regardless of the diagnosis at readmission.
Number of participants who are admitted to the intensive care unit after the operation. | Day 30
  Admission to the intensive care unit after the operation.
Number of patients in need of re-operation | Day 30
  Need for re-operation due to complications

OTHER OUTCOMES:
Percentage of staff who have received training | This outcome will be evaluated from when the implementation period starts and until it finishes. The length of this period is 6 months. Staff participation in the training will be registred, and the sessions repeated during the 6 months.
  It will be registered how many of the staff have received the training, the target being 80%. Staff participation in the training will be registred, and the sessions repeated during the 6 months, until 80% of the staff, or more, have recieved the training.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyhoff, MD, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark